CLINICAL TRIAL: NCT02839200
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Active-reference, Parallel-group, Polysomnography Dose-response Study to Assess the Efficacy and Safety of ACT-541468 in Adult Subjects With Insomnia Disorder
Brief Title: Efficacy and Safety of ACT-541468 in Adult Subjects With Insomnia Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-078A201
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Insomnia Disorder
Keywords: Insomnia; Polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ACT-541468 5 mg (Experimental): Each subject receives one 5-mg ACT-541468 capusle (+ one placebo capsule), once daily in the evening for 4 weeks
  Interventions: Drug: ACT-541468 5 mg; Drug: Placebo 1
- ACT-541468 10 mg (Experimental): Each subject receives one 10-mg ACT-541468 capusle (+ one placebo capsule), once daily in the evening for 4 weeks
  Interventions: Drug: ACT-541468 10 mg; Drug: Placebo 1
- ACT-541468 25 mg (Experimental): Each subject receives one 25-mg ACT-541468 capsule (+ one placebo capsule), once daily in the evening) for 4 weeks
  Interventions: Drug: ACT-541468 25 mg; Drug: Placebo 1
- ACT-541468 50 mg (Experimental): Each subject receives two 25-mg ACT-541468 capsules, once daily in the evening for 4 weeks
  Interventions: Drug: ACT-541468 25 mg
- Zolpidem (Active Comparator): Each subject receives one 10-mg zolpidem capsule (+ one placebo capusle), once daily in the evening for 4 weeks
  Interventions: Drug: Zolpidem; Drug: Placebo 2
- Placebo (Placebo Comparator): Each subject receives two placebo capsules, once daily in the evening for 4 weeks
  Interventions: Drug: Placebo 1

INTERVENTIONS:
Drug: ACT-541468 5 mg — Capsule for oral administration containing ACT-541468 at a strength of 5 mg
  Arms: ACT-541468 5 mg
Drug: ACT-541468 10 mg — Capsule for oral administration containing ACT-541468 at a strength of 10 mg
  Arms: ACT-541468 10 mg
Drug: ACT-541468 25 mg — Capsule for oral administration containing ACT-541468 at a strength of 25 mg
  Arms: ACT-541468 25 mg; ACT-541468 50 mg
Drug: Zolpidem — Over-encapsulated zolpidem tablet at a strength of 10 mg
  Arms: Zolpidem
Drug: Placebo 1 — Placebo capsules matching ACT-541468 capsules
  Arms: ACT-541468 10 mg; ACT-541468 25 mg; ACT-541468 5 mg; Placebo
Drug: Placebo 2 — Placebo capsules matching over-encapsulated zolpidem
  Arms: Zolpidem

SUMMARY:
This study evaluates the dose response of ACT-541468 on the change of WASO from baseline to Days 1 and 2, assessed by PSG.

DETAILED DESCRIPTION:
This study consists of the following phases: screening phase; double-blind treatment phase; safety follow-up phase. Safety is monitored throughout the study.

ELIGIBILITY:
Principal inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male or female aged 18-64 years (inclusive).
* Women of childbearing potential must have negative pregnancy tests and use reliable methods of contraception up to 30 days after EOT.
* Body mass index (BMI): 18.5 ≤ BMI (kg/m2) < 32.0.
* Insomnia disorder according to DSM-5 criteria.
* Insufficient sleep quantity as collected subjectively in the sleep diary and validated objectively by polysomnography.
* Insomnia Severity Index score ≥ 15.

Principal exclusion Criteria:

* Any current history of sleep disorder other than insomnia, or any lifetime history of related breathing disorder, periodic limb movement disorder, restless legs syndrome, circadian rhythm disorder, rapid eye movement (REM) behavior disorder, or narcolepsy.
* Self-reported usual daytime napping ≥ 1 hour per day, and ≥ 3 days per week.
* Caffeine consumption ≥ 600 mg per day.
* Shift work within 2 weeks prior to the screening visit, or planned shift work during study.
* Travel ≥ 3 time zones within 1 week prior to the screening visit, or planned travel > or= 3 time zones during study.
* Hematology or biochemistry test results deviating from the normal range to a clinically relevant extent as per judgment of the Investigator.
* AST and/or ALT > 2 × ULN and/or direct bilirubin > 1.5 × ULN (except known history of Gilbert's syndrome).
* Severe renal impairment (known or defined as estimated creatinine clearance < 30 mL/min).
* History or clinical evidence of any disease or medical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the study assessments.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (30):
- United States (15):
  - Investigator Site, Santa Monica, California
  - Investigator Site, Upland, California
  - Investigator Site, Brandon, Florida
  - Investigator Site, Clearwater, Florida
  - Investigator Site, Coral Gables, Florida
  - Investigator Site, DeLand, Florida
  - Investigator Site, Hollywood, Florida
  - Investigator Site, Miami, Florida
  - Investigator Site, Atlanta, Georgia
  - Investigator Site, Chicago, Illinois
  - Investigator Site, Indianapolis, Indiana
  - Investigator Site, Novi, Michigan
  - Investigator Site, Las Vegas, Nevada
  - Investigator Site, New York, New York
  - Investigator Site, Cincinnati, Ohio
- Germany (5):
  - Investigator Site, Berlin
  - Investigator Site, Dresden
  - Investigator Site, Hamburg
  - Investigator Site, Hanover
  - Investigator Site, Schwerin
- Hungary (3):
  - Investigator Site, Budapest
  - Investigator Site, Szeged
  - Investigator Site, Törökbálint
- Israel (2):
  - Investigator Site, Beersheba
  - Investigator Site, Haifa
- Spain (3):
  - Investigator Site, Barcelona
  - Investigator Site, Madrid
  - Investigator Site, Zaragoza
- Sweden (2):
  - Investigator Site, Gothenburg
  - Investigator Site, Örebro

REFERENCES:
- [Derived] Dutta S, Singhal S, Shah R, Charan J, Dhingra S, Haque M. Daridorexant as a novel pharmacotherapeutic approach in insomnia: a systematic review and meta-analysis. Expert Opin Drug Saf. 2023 Jul-Dec;22(12):1237-1251. doi: 10.1080/14740338.2023.2243217. Epub 2023 Aug 7. PMID 37526060
- [Derived] Di Marco T, Scammell TE, Meinel M, Seboek Kinter D, Datta AN, Zammit G, Dauvilliers Y. Number, Duration, and Distribution of Wake Bouts in Patients with Insomnia Disorder: Effect of Daridorexant and Zolpidem. CNS Drugs. 2023 Jul;37(7):639-653. doi: 10.1007/s40263-023-01020-9. Epub 2023 Jul 21. PMID 37477771
- [Derived] Dauvilliers Y, Zammit G, Fietze I, Mayleben D, Seboek Kinter D, Pain S, Hedner J. Daridorexant, a New Dual Orexin Receptor Antagonist to Treat Insomnia Disorder. Ann Neurol. 2020 Mar;87(3):347-356. doi: 10.1002/ana.25680. Epub 2020 Feb 5. PMID 31953863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 38 sites in 6 countries (Germany, Hungary, Israel, Spain, Sweden, and the USA)
Pre-assignment Details: Screening details: screening period (screening visit followed by at least 7 days at home) and a run-in period (2 PSG nights on single-blind placebo, followed by 5-12 days with no treatment), and lasting a max. of 28 days. N = 360 subjects were randomized; N = 359 subjects were treated; N = 1 subject discontinued due to "randomization error".
Groups:
- ACT-541468 5 mg: Each subject received one 5-mg ACT-541468 capusle (+ one placebo capsule), once daily in the evening for 4 weeks
  ACT-541468 5 mg: Capsule for oral administration containing ACT-541468 at a strength of 5 mg
  Placebo 1: Placebo capsules matching ACT-541468 capsules
- ACT-541468 10 mg: Each subject received one 10-mg ACT-541468 capusle (+ one placebo capsule), once daily in the evening for 4 weeks
  ACT-541468 10 mg: Capsule for oral administration containing ACT-541468 at a strength of 10 mg
  Placebo 1: Placebo capsules matching ACT-541468 capsules
- ACT-541468 25 mg: Each subject received one 25-mg ACT-541468 capsule (+ one placebo capsule), once daily in the evening for 4 weeks
  ACT-541468 25 mg: Capsule for oral administration containing ACT-541468 at a strength of 25 mg
  Placebo 1: Placebo capsules matching ACT-541468 capsules
- ACT-541468 50 mg: Each subject received two 25-mg ACT-541468 capsules, once daily in the evening for 4 weeks
  ACT-541468 25 mg: Capsule for oral administration containing ACT-541468 at a strength of 25 mg
- Zolpidem: Each subject received one 10-mg zolpidem capsule (+ one placebo capusle), once daily in the evening for 4 weeks
  Zolpidem: Over-encapsulated zolpidem tablet at a strength of 10 mg
  Placebo 2: Placebo capsules matching over-encapsulated zolpidem
- Placebo: Each subject received two placebo capsules, once daily in the evening for 4 weeks
  Placebo 1: Placebo capsules matching ACT-541468 capsules
Period: Overall Study
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Zolpidem | Placebo
Started | 60 | 59 | 60 | 61 | 60 | 60
Completed | 56 | 58 | 59 | 61 | 58 | 59
Not Completed | 4 | 1 | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Randomized in error | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ACT-541468 25 mg: Each subject received one 25-mg ACT-541468 capsule (+ one placebo capsule), once daily in the evening) for 4 weeks
  ACT-541468 25 mg: Capsule for oral administration containing ACT-541468 at a strength of 25 mg
  Placebo 1: Placebo capsules matching ACT-541468 capsules
- Total: Total of all reporting groups
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Zolpidem | Placebo | Total
Number analyzed (Participants) | 60 | 58 | 60 | 61 | 60 | 60 | 359
Age, Continuous [Median (Full Range); unit: years] | 41 [22 to 64] | 48 [21 to 63] | 48 [18 to 64] | 46 [18 to 63] | 43 [23 to 61] | 48 [23 to 64] | 47 [18 to 64]
Age, Customized [Count of Participants; unit: Participants] — Age categorical (Unit: subjects)
  Participants
    Adults (18-64 years) | 60 | 58 | 60 | 61 | 60 | 60 | 359
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 39 | 39 | 38 | 38 | 230
  Male | 22 | 20 | 21 | 22 | 22 | 22 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 9 | 5 | 4 | 9 | 39
  Not Hispanic or Latino | 51 | 54 | 51 | 56 | 56 | 51 | 319
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 5 | 8 | 4 | 5 | 6 | 7 | 35
  White | 54 | 49 | 56 | 56 | 54 | 52 | 321
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Wake After Sleep Onset (WASO) From Baseline to Days 1 and 2
Description: WASO is the time in minutes spent awake after onset of persistent sleep until lights on as determined by polysomnography (PSG)
Time Frame: Baseline and Days 1&2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Zolpidem | Placebo
Number analyzed (Participants) | 60 | 58 | 60 | 61 | 60 | 60
minutes | -28.4 (4.24) | -32.3 (4.32) | -37.7 (4.25) | -47.1 (4.21) | -29.9 (4.30) | -21.4 (4.24)
Statistical Analysis 1: Comparison: ACT-541468 5 mg vs ACT-541468 10 mg vs ACT-541468 25 mg vs ACT-541468 50 mg vs Placebo; Multiple Comparison Procedure-Modeling (MCP-Mod) was used to assess a dose-response across placebo and all ACT-541468 doses. The null hypothesis of "no dose-response" was rejected if at least one of the six Multiple Contrasts Tests (MCTs) had a multiplicity adjusted p-value <0.05. The analysis was performed using the R-package "DoseFinding" (Bornkamp B, Pinheiro J, Bretz F. Planning and analyzing dose finding experiments. 2016. Available from: cranrprojects.org/web/packages/DoseFinding.); Test type: Other; p < 0.001, Multiple Comparison Procedure-Model
Statistical Analysis 2: Comparison: ACT-541468 5 mg vs Placebo; Test type: Other; p = 0.241, ANCOVA; LS mean difference = -7, 95% CI 2-sided [-18.7 to 4.7], Standard Error of Mean 5.95 — Parameter Dispersion Type and Dispersion Value: Standard error of the LS mean
Statistical Analysis 3: Comparison: ACT-541468 10 mg vs Placebo; Test type: Other; p = 0.072, ANCOVA; LS Mean difference = -10.8, 95% CI 2-sided [-22.6 to 1], Standard Error of Mean 6 — Parameter Dispersion Type and Dispersion Value: Standard error of the LS mean
Statistical Analysis 4: Comparison: ACT-541468 25 mg vs Placebo; Test type: Other; p = 0.007, ANCOVA; LS Mean difference = -16.2, 95% CI 2-sided [-27.9 to -4.5], Standard Error of Mean 5.95 — Parameter Dispersion Type and Dispersion Value: Standard error of the LS mean
Statistical Analysis 5: Comparison: ACT-541468 50 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; LS Mean difference = -25.6, 95% CI 2-sided [-37.3 to -13.9], Standard Error of Mean 5.92 — Parameter Dispersion Type and Dispersion Value: Standard error of the LS mean
Statistical Analysis 6: Comparison: Zolpidem vs Placebo; Test type: Other; p = 0.155, ANCOVA; LS Mean difference = -8.5, 95% CI 2-sided [-20.4 to 3.3], Standard Error of Mean 5.97 — Parameter Dispersion Type and Dispersion Value: Standard error of the LS mean

2. Secondary Outcome: Change in Latency to Persistent Sleep (LPS) From Baseline to Days 1 and 2
Description: LPS is the duration of time in minutes from lights off to persistent sleep onset as determined by PSG
Time Frame: Baseline and Days 1&2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Zolpidem | Placebo
Number analyzed (Participants) | 60 | 58 | 60 | 61 | 60 | 60
Minutes | -26.88 (45.42) | -29.31 (26.79) | -36.14 (34.34) | -36.41 (26.71) | -45.14 (32.82) | -22.02 (46.63)

3. Secondary Outcome: Change in Subjective Latency to Sleep Onset (sLSO) From Baseline to Week 4
Description: sLSO is the self-reported time to fall asleep, as reported in the sleep diary
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Zolpidem | Placebo
Number analyzed (Participants) | 60 | 58 | 60 | 61 | 60 | 60
Minutes | -13.38 (27.79) | -21.07 (24.26) | -15.50 (25.51) | -23.65 (24.12) | -19.98 (19.28) | -16.32 (21.16)

4. Secondary Outcome: Change in Subjective Wake After Sleep Onset (sWASO) From Baseline to Week 4
Description: sWASO is the self-reported time spent awake after sleep onset as reported in the sleep diary.
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Zolpidem | Placebo
Number analyzed (Participants) | 51 | 45 | 53 | 49 | 48 | 50
Minutes | -31.32 (33.32) | -24.35 (33.4) | -29.8 (39.88) | -35.45 (37.53) | -29.08 (27.28) | -23.61 (32.62)

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected from Screening to Safety Follow-up period. Below, data are reported for treatment-emergent adverse events (TEAEs).
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Zolpidem | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58 | 0/60 | 0/61 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 2/58 | 0/60 | 1/61 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 21/60 | 22/58 | 23/60 | 21/61 | 24/60 | 18/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT-541468 5 mg (N=60) | ACT-541468 10 mg (N=58) | ACT-541468 25 mg (N=60) | ACT-541468 50 mg (N=61) | Zolpidem (N=60) | Placebo (N=60)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT-541468 5 mg (N=60) | ACT-541468 10 mg (N=58) | ACT-541468 25 mg (N=60) | ACT-541468 50 mg (N=61) | Zolpidem (N=60) | Placebo (N=60)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chromatopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces pale (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (5) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 4 (5) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 4 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ECG signs of myocardial infarction (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 5 (5) | 5 (5) | 5 (6) | 6 (8) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 3 (4) | 3 (3) | 4 (5) | 4 (5) | 3 (3) | 3 (3)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT02839200/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT02839200/SAP_001.pdf